CLINICAL TRIAL: NCT03961594
Title: Evaluation of New Hemodynamic Indices to Predict Response to Volemic Expansion in Septic Shock
Brief Title: Evaluation of New Hemodynamic Indices
Acronym: EVOLVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: '2018-38'; 2018-A01078-47 (Registry Identifier: APHM)
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Intervention Model Description: Inclusions will be based on the formal preliminary indication of a volume expansion test to avoid over inclusions and side effects of an undesired volume expansion.
  The collection of data is done in daily practice, relies on routine care and does not require additional devices
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- volume expansion in the ventilated patient (Other): Including 51 patients, ventilated, under vasopressors suffering from septic shock. GLS, cardiac output, VVP, VVE, blood pressure, Eadyn, EtCO2 will be measured before and after ELJP. In the event of an increase of more than 10% in cardiac output during the ELJP, patients will receive a volume expansion of 500ml of balanced crystalloids. The same measurements will be repeated immediately at the end of the volume expansion and 20 minutes after the end of the infusion. Patients with a 15% increase in cardiac output at the end of volume expansion will be classified as responders. Patients with a 15% increase in cardiac output 20minutes after the end of volume expansion will be classified as persistent responders.
  Interventions: Other: expansion volémique

INTERVENTIONS:
Other: expansion volémique — cardiac output, VVP, VVE, blood pressure, Eadyn, EtCO2 will be measured before and after ELJP. In the event of an increase of more than 10% in cardiac output during the ELJP, patients will receive a volume expansion of 500ml of balanced crystalloids. The same measurements will be repeated immediately at the end of the volume expansion and 20 minutes after the end of the infusion. Patients with a 15% increase in cardiac output at the end of volume expansion will be classified as responders.

SUMMARY:
The objective is to determine the sensitivity and specificity via Receiver Operating Characteristic (ROC) curve of Global Longitudinal Strain (GLS) The secondary objectives are the same for the change in the amount of carbon dioxide exhaled (ΔEtCO2) and dynamic arterial elastance (Eadyn). it will also determine the sensitivity and specificity of these indices, either individually or combined to determine persistent responders to volemic expansion.

DETAILED DESCRIPTION:
The best practice recommendations are to evaluate the preload dependence before performing a vascular filling test. This evaluation is based on the analysis of dynamic hemodynamic indices such as the variation of pulsed pressure (VPP), the variation of the volume of ejection (VVE) or the variation of the cardiac output during the realization of a test of rising of passive leg (ELJP). However, these indices require strict validation conditions.

New hemodynamic indices have appeared recently and appear promising in the evaluation of preload dependence. Among them, the analysis of longitudinal myocardial deformity by speckle tracking (GLS) and its variation during an ELJP (ΔGLS). The analysis of changes in the amount of CO2 exhaled (ΔEtCO2) reflects cardiac output in ventilated patients or the analysis of dynamic arterial elastance (Eadyn) calculated by comparing the VPP and the EVV which is a reflection of the coupling between the left ventricle and the arterial network.

In this work the assumption that the analysis of Δ GLS, ΔEtCO2 and Eadyn can predict the response to volume expansion in the ventilated patient, in septic shock under vasopressor.

The investigators include at least 51 patients, ventilated, under vasopressors with septic shock. GLS, cardiac output, VVP, VVE, blood pressure, Eadyn, EtCO2 will be measured before and after ELJP. In the event of an increase of more than 10% in cardiac output during the ELJP, patients will receive a volume expansion of 500ml of balanced crystalloids. The same measurements will be repeated immediately at the end of the volume expansion and 20 minutes after the end of the infusion. Patients with a 15% increase in cardiac output at the end of volume expansion will be classified as responders. Patients with a 15% increase in cardiac output 20minutes after the end of volume expansion will be classified as persistent responders.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting a shock whose etiology is considered as septic.
* Patient whose hemodynamic state justifies the infusion of vasopressor.
* Patient monitored by a cardiac output measurement system calibrated by transpulmonary thermodilution.
* Intubated patient with expired capnia monitoring
* Patient with signs of low cardiac output

Exclusion Criteria:

* Patient with a contraindication in the leg lift test.
* Patient with abdominal compartment syndrome.
* Patient with amputation of one or both lower limbs.
* Pregnant woman eliminated by a systematic pregnancy test at the entrance to the intensive care unit.
* Minor patient.
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2018-07-19 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Passive leg lift test (ELJP) | 20 minutes
  The ELJP consists of a tilting maneuver of the patient's bed from a proclive position at 30 ° to a 0 ° chest position and limbs less than 30 °. This maneuver allows the recruitment of venous blood contained in the lower limbs to the heart and to "mimic" a test of volemic expansion and its hemodynamic repercussions. This maneuver is widely described in the literature for this indication and does not involve any particular risk for the patient. The measurements are made at 1 minute of the end of the tilting (chest at 0 °). The maneuver lasts 1min30 before returning the patient to his initial position

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France